CLINICAL TRIAL: NCT00895206
Title: Individually Adapted Immunosuppression in de Novo Renal Transplantation Based on Immune Function Monitoring: a Prospective Randomised Study
Acronym: CD4-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/640
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): individual adapted immunosuppression
  Interventions: Drug: individual adapted immunosuppression
- 2 (Active Comparator): golden standard therapy
  Interventions: Drug: golden standard therapy

INTERVENTIONS:
Drug: individual adapted immunosuppression — individual adapted immunosuppression
  Arms: 1
Drug: golden standard therapy — golden standard therapy
  Arms: 2

SUMMARY:
This study is an open, randomised trial in which one group of patients (control) will receive the golden standard therapy and the other group (treatment) will receive individually adapted immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* First or second kidney transplantation
* Males and females, 18 years old or older
* Women of childbearing potential must have a negative serum or urine pregnancy test with sensitivity equal to at least 50 mIU/mL
* Patients must be capable of understanding the purpose and risks of the study and must sign an informed consent form

Exclusion Criteria:

* Multiple organ transplantation (eg. kidney-pancreas, kidney-heart, kidney-liver,...)
* Transplantation of a patient who received another organ transplant previously except one kidney transplant
* Recipients of HLA-identical living-related renal transplants
* Patients with PRA > 10%, patients who have lost a first graft from rejection.
* Pregnant or lactating women
* WBC =< 2.5 x 109/L (IU), platelet count =< 100 x 109/L (IU), or Hb =< 6g/dl at the time of entry into the study
* Active peptic ulcer
* Severe diarrhea or other gastrointestinal disorders which might interfere with the ability to absorb oral medication, including diabetic patients with previously diagnosed diabetic gastroenteropathy
* Known HIV-1 or HTLV-1 positive tests
* History of malignancy in the past 5 years (with the exception of adequately treated basal or squamous skin cell carcinoma)
* The use of investigational drugs or other immunosuppressive drugs as those specified in this protocol
* Patients receiving bile acid sequestrants
* Psychological illness or condition interfering with the patient's compliance or ability to understand the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-05; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Graft function as measured by Cr EDTA AUC | at 1 year

SECONDARY OUTCOMES:
Graft survival | at 1 year
Patient survival | at 1 year
Graft function measured by estimated GFR (eGFR) (MDRD and Cockroft-Gault) | at 1 year
Frequency of biopsy proven acute rejection episodes | at 1 year
Incidence of biopsy proven acute rejection (BPAR) and clinical (non-biopsy proven) acute rejection episodes treated by a full course anti-rejection therapy (e.g. steroids) (Treatment of rejection according to center practice). | at 1 year
Incidence of rejection treated by antibodies (OKT3, ATG) | at 1 year
Time to first rejection (days) | at 1 year
Severity of rejection as assessed by BANFF 2005 score | at 1 year
Number of acute rejections per patient | at 1 year
Plasma creatinine and eGFR | at month 1, 3 and yearly (2 and 3 years)
Measured GFR | at month 3 and yearly
Proteinuria | at month 1, 3 and at 1 and 3 years
Incidence and score of borderline changes and acute rejection | in month 3 and month 12 biopsy
Incidence and score of chronic alloimmune injury/rejection and nonimmune injury | in month 3 and month 12 biopsies (BANFF 2005)
Development and evolution of glucose abnormalities | at 1 year
blood pressure | at 1 year
ambulatory 24-hr blood pressure monitoring | at 1 year and 3 years
Left ventricular mass assessed by echocardiography | at 1 year and 3 years
Fasting lipid profile | at baseline, month 1,3,6 and yearly
CMV infection (as measured with whole blood PCR) and disease | at 1 year
Polyoma virus replication as measured by whole blood PCR | at 1 year
Incidence of BK nephritis | in month 3 and month 12 biopsies
Incidence of PTLD and Nonmelanoma skin cancer | at 1 year and yearly
Incidence of EBV reactivation (as measured with whole blood PCR) | at 1 year and yearly

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be